CLINICAL TRIAL: NCT02534922
Title: Phase I Open-Label, Dose-Escalation and Pharmacokinetic Study of Subcutaneous Prolanta™ in Subjects With Recurrent or Persistent Epithelial Ovarian Cancer, Primary Peritoneal Cancer, or Fallopian Tube Cancer
Brief Title: Study of Prolanta™ in Recurrent or Persistent Epithelial Ovarian Cancer
Acronym: ProlantaOC
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oncolix, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONC-OC-001
Record Dates: First submitted 2015-08-24; First posted 2015-08-28 (Estimated); Last update posted 2018-02-14 (Actual); Status verified 2018-02

CONDITIONS: Ovarian Cancer; Peritoneal Cancer; Fallopian Tube Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Daily dosing (Experimental): Daily subcutaneous dosing of Prolanta, a human prolactin receptor antagonist
  Interventions: Biological: Prolanta, a human prolactin receptor antagonist

INTERVENTIONS:
Biological: Prolanta, a human prolactin receptor antagonist — Daily subcutaneous dosing

SUMMARY:
This trial is a Phase I open-label safety study of Prolanta™, a recombinant analog of the human prolactin protein with a single amino acid substitution to create an antagonist of the prolactin receptor. The Sponsor believes that blocking the prolactin receptor in patients with ovarian and other cancers will be effective as a monotherapy or in combination with other chemotherapies. This Phase I study will be conducted in Subjects with recurrent or persistent epithelial ovarian cancer, primary peritoneal cancer, or fallopian tube cancer.

DETAILED DESCRIPTION:
This study is a first-in-human study designed to establish preliminary human safety, tolerability and pharmacokinetic parameters of Prolanta monotherapy in patients with recurrent or persistent ovarian cancer, primary peritoneal cancer, or fallopian tube cancer. In addition, biomarkers related to the activity of human prolactin will be examined in tumor samples obtained prior to treatment and at the end of study treatment to determine the pharmacodynamics of the dose levels of Prolanta administered. Three dosing levels will be evaluated, and the dose at which no dose-limiting toxicities are observed will be the recommended Phase II dose.

Because of its antagonist effect and the expected lower toxicity, Sponsor believes that Prolanta may be administered continuously as a monotherapy or in conjunction with the periodic administration of chemotherapy (i.e., a dual therapy). The dosing schedule to be used in this trial is designed to evaluate, in increments, the safety and tolerability of Prolanta over this 90 day cycle. Subjects will be assessed for antibody presence throughout the study, initially on a weekly basis and then bi-weekly. Subjects will be initially dosed for 28 days followed by a safety assessment period, and then continue for an additional 56 days if no toxicities are observed.

The primary objectives of this study are to determine the safety and tolerability of Prolanta in women with recurrent ovarian cancer and to determine the optimal dose of Prolanta to use in Phase II studies. The safety evaluation will be determined by assessing treatment-emergent adverse events, physical examination, ECG, changes in clinical laboratory results including clinical chemistry, hematology and urinalysis, changes in pituitary hormone levels, and vital signs including blood pressure, pulse and respiratory rate. The optimal dose of Prolanta will be determined by evaluating both the safety profile and blood levels of Prolanta. If possible, the effect of the Prolanta dose on tumor biomarkers and tumor burden will also be used to determine the optimally bioactive Phase II dose level.

The secondary objectives of this study are (i) to determine the pharmacokinetic parameters of Prolanta including Cmax, Tmax, half-life and area under the curve (AUC); (ii) to determine the effect of treatment with Prolanta on tumor markers; (iii) to determine clinical efficacy of Prolanta by Response Evaluation Criteria in Solid Tumors (RECIST), version 1.1

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have recurrent or persistent epithelial ovarian cancer, primary peritoneal cancer or fallopian tube cancer. Histologic confirmation of the original primary tumor is required.
* Subjects shall have had cytoreductive (debulking) surgery.
* Formalin-fixed, paraffin-embedded tumor tissue blocks must be available for each Subject upon enrollment and provided to Sponsor within 7 days of Day 1.
* Subjects must have measurable and accessible disease.
* Subjects must either: (i) have relapsed within 6 months after (or progressed during) their last platinum regimen (this may be their primary/ adjuvant regimen); or (ii) have progressed after 2 or more prior platinum regimens (regardless of duration since most recent platinum regimen); or (iii) can not tolerate platinum therapy due to hypersensitivity or other allergic reactions.
* In addition to the first platinum-based chemotherapy, Subjects are allowed to have previously received no more than two additional cytotoxic regimens for management of recurrent or persistent disease. "Cytotoxic regimens" include any agent that targets the genetic and/or mitotic apparatus of dividing cells, resulting in dose-limiting toxicity to the bone marrow and/or gastrointestinal mucosa.
* Resolution of any effects of prior therapy (except alopecia) to NCI CTCAE v4.03 grade ≤2 and to baseline laboratory values as defined in inclusion criteria #14.
* Eastern Cooperative Oncology Group (ECOG) performance status: 0 - 2
* Life expectancy >12 weeks
* Any hormonal therapy directed at the malignant tumor must be discontinued at least one week prior to registration. Continuation of hormone replacement therapy is permitted.
* Any prior therapy directed at the malignant tumor, including immunologic agents and chemotherapy, must be discontinued at least four weeks prior to registration (6 weeks for nitrosoureas or mitomycin C).
* Patients must have normal organ and marrow function as defined.
* Normal electrocardiogram (ECG) with corrected QT interval (QTc) ≤470 msec.

Exclusion Criteria:

* Currently receiving any other investigational agents or having participated in an investigational therapy trial within 30 days.
* Planned pregnancy, currently pregnant or breastfeeding.
* Females of childbearing potential who are not using a medically accepted means of contraception (e.g., intrauterine device, oral contraceptive, implant, Depo-Provera®, or barrier devices with spermicide) when engaging in sexual intercourse.
* History or evidence upon physical examination of central nervous system (CNS) disease, including primary brain tumor, seizures not controlled with standard medical therapy, any brain metastases or history of cerebrovascular accident, transient ischemic attack or subarachnoid hemorrhage within 6 months of registration on this study.
* Serious pre-existing medical conditions such as severe heart disease or uncontrolled: infections, hypertension, hypercalcemia, diabetes, or psychogenic disorders.
* Have any other concurrent malignancies, except adequately treated in situ carcinoma of the cervix or basal cell or squamous cell carcinoma of the skin. (Subjects who have undergone potentially curative therapy for a prior malignancy are eligible provided there is no evidence of disease for ≥ 5 years and patient is deemed to be at low risk for recurrence.)
* Any other significant medical condition that, in the opinion of the Investigator, would significantly decrease study compliance, jeopardizes the safety of the patient, or affects the validity of the trial results.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2016-02; Primary Completion 2019-02 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Number of Subjects with Treatment Related Adverse Events by CTCAE v4.03 | 90 days
  The Common Toxicity Criteria for Adverse Effects (CTCAE), version 4.03, graded toxicity scale will be utilized to assess local and systemic toxicity. Dose Limiting Toxicity is defined as any grade 3 or higher toxicity or any grade 2 hypersensitivity reaction or neurologic toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Michael T Redman, Study Director — Oncolix, Inc.
Locations (1):
- ITOR/GHS, Greenville, South Carolina, United States